CLINICAL TRIAL: NCT01495923
Title: Randomized, Double-blind, Comparative-effectiveness Study Comparing Epidural Steroid Injections to Gabapentin in Patients With Lumbosacral Radiculopathy
Brief Title: Steroids Versus Gabapentin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); Brooke Army Medical Center (U.S. Federal Agency); Landstuhl Regional Medical Center (U.S. Federal Agency); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency); Case Western Reserve University (Other); Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Steven P. Cohen, Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00047152
Record Dates: First submitted 2011-12-15; First posted 2011-12-20 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Sciatica; Radiculopathy
Keywords: low back pain; radiculopathy; injection
MeSH Terms: conditions — Sciatica; Radiculopathy; Low Back Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural steroids (Experimental): Injection of steroids into the epidural space
  Interventions: Procedure: epidural steroid injection; Drug: Placebo gabapentin
- Gabapentin (Active Comparator): Titration of gabapentin to effect
  Interventions: Procedure: Sham epidural steroid injection; Drug: Gabapentin

INTERVENTIONS:
Procedure: epidural steroid injection — Injection of steroids and local anesthetic into the epidural space
  Arms: Epidural steroids
Procedure: Sham epidural steroid injection — Injection of saline into the back muscles
  Arms: Gabapentin
Drug: Gabapentin — Titration of gabapentin to effect
  Arms: Gabapentin
Drug: Placebo gabapentin — Titration of placebo gabapentin
  Arms: Epidural steroids

SUMMARY:
The purpose of this study is to determine whether pharmacotherapy or epidural steroid injections are a better treatment for lumbosacral radicular pain.

142 patients referred to a participating pain clinic with lumbosacral radiculopathy will be randomized in a 1:1 ratio to receive one of two treatments. Half (n=71) of the patients will be allocated to receive an epidural steroid injection (ESI; group I), with an equal number allocated to receive gabapentin (group II). Patients & evaluating physicians will be blinded. Follow-up will be through 3-months after treatment.

DETAILED DESCRIPTION:
142 patients referred to a participating pain clinic with lumbosacral radiculopathy will be randomized in a 1:1 ratio to receive one of two treatments. Half (n=71) of the patients will be allocated to receive an ESI (group I), with an equal number allocated to receive gabapentin (group II).

Group I patients with unilateral symptoms will receive (unilateral) transforaminal ESI, while those with bilateral symptoms will receive (central) interlaminar ESI, as is common practice.

In group II patients who receive gabapentin, the dose will be titrated to between 1800 mg/d and 2700 mg/d in TID dosing, but may be lowered or elevated (up to 3600 mg/d) depending on the clinical circumstances. To ensure blinding, these patients will also receive midline (for patients with bilateral symptoms who would receive interlaminar ESI) or unilateral paraspinal (for patients with unilateral symptoms who would receive transforaminal ESI) normal saline into the interspinal ligaments or paraspinal musculature, respectively. Injections and medication titration will commence on the same day.

Rescue medications will consist of tramadol 50 mg 1 to 2 tablets every 6 hours PRN (up to 8/d) and/or ibuprofen 400-800 mg every 6 hours PRN (not-to-exceed 3000 mg/d). Patients already taking analgesics, including opioids, can continue on these medications "as needed".

The first follow-up visit will be scheduled 1-month from the start of treatment. A positive outcome will be defined as a > 2-point decrease in leg pain coupled with a positive satisfaction rating. Subjects who obtain a positive outcome at their initial 1-month follow-up visit will remain in the study and return for the final 3-month follow-up visit. Those with a negative outcome will exit the study "per protocol" to receive standard care, which may consist of unblinded ESI, medical management with drugs such as gabapentin (for those who did not receive gabapentin) and antidepressants, and physical therapy. Subjects who obtain a positive outcome at 1-month but experience a recurrence before their 3-month follow-up visit will also exit the study per protocol, with their final outcome measures recorded before they receive standard care. At all follow-up visits, pill counts will be conducted to determine medication compliance.

ELIGIBILITY:
Inclusion Criteria:

* Lumbosacral radicular pain based on history and physical exam (e.g. pain radiating into one or both lower extremities, sensory loss, muscle weakness, positive straight leg raising test etc.)
* Numerical Rating Scale leg pain score > 4 (or if 3/10, greater or equal to back pain)
* MRI evidence of spinal pathology consistent with symptoms

Exclusion Criteria:

* Untreated coagulopathy
* Previous spine surgery
* No MRI study
* Leg pain > 4 years duration Epidural steroid injection within past 3 years Cauda equina syndrome Previous failed trials with gabapentin or pregabalin Allergic reactions to gabapentin or pregabalin Referrals from surgery for diagnostic injections for surgical evaluation Serious medical or psychiatric that condition that might preclude optimal outcome or interfere with participation, such as the need for uninterrupted anticoagulation.

Pregnancy

Ages: 17 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (3):
- United States (3):
  - Naval Hospital-San Diego, San Diego, California
  - Johns Hopkins, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland

REFERENCES:
- [Derived] Cohen SP, Hanling S, Bicket MC, White RL, Veizi E, Kurihara C, Zhao Z, Hayek S, Guthmiller KB, Griffith SR, Gordin V, White MA, Vorobeychik Y, Pasquina PF. Epidural steroid injections compared with gabapentin for lumbosacral radicular pain: multicenter randomized double blind comparative efficacy study. BMJ. 2015 Apr 16;350:h1748. doi: 10.1136/bmj.h1748. PMID 25883095

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 15, 2011 and June 10, 2014 145 participants were recruited at 8 sites. The sites included 4 joint service military treatment facilities, 3 of which serve as teaching hospitals and 1 of which is located in Europe; a Veteran's Administration hospital; and 3 civilian teaching hospitals.
Groups:
- Epidural Steroid Injection: If randomized to this group, participants received either a transforaminal injection for unilateral pain or an interlaminar injection for bilateral pain and placebo medication. The level and type of injection to be given was determined by signs, symptoms, and radiological findings.
- Gabapentin: If randomized to this group participants received gabapentin medication and a placebo intramuscular injection. The gabapentin was uptitrated to a therapeutic dose using a titration schedule.
Period: Overall Study
Arm/Group | Epidural Steroid Injection | Gabapentin
Started | 73 | 72
Completed | 73 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Epidural Steriod Injections: Participants that had lumbosacral radicular pain secondary to herniated disc or spinal stenosis who receive a real epidural steroid injection and placebo medication as treatment.
- Gabapentin: Participants that had lumbosacral radicular pain secondary to herniated disc or spinal stenosis who receive real gabapentin and a placebo injection as treatment.
- Total: Total of all reporting groups
Arm/Group | Epidural Steriod Injections | Gabapentin | Total
Number analyzed (Participants) | 73 | 72 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 72 | 145
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (14) | 41.7 (11.9) | 42.7 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 13 | 38
  Male | 48 | 59 | 107
Region of Enrollment [Number; unit: participants]
  United States | 67 | 67 | 134
  Germany | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Average Leg Pain at 1 Month Measured Using the Numeric Pain Scale
Description: This outcome measure compares the average leg pain at baseline to the average leg pain 1 month after the start of treatment. This is measured using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0-10. 0 being no pain at all and 10 being the worst imaginable pain possible. The epidural steroid injection group is compared to the gabapentin group.
Time Frame: 1 month after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Epidural Steroid Injection: This group received an epidural steroid injection and placebo medication.
- Gabapentin: This group received gabapentin medication and a placebo injection.
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 73 | 72
units on a scale | 3.3 (2.6) | 3.7 (2.6)

2. Primary Outcome: Average Leg Pain at 3 Months Measured Using the Numeric Pain Scale
Description: This outcome measure compares the average leg pain at baseline to the average leg pain 3 month after the start of treatment. This is measured using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0-10. 0 being no pain at all and 10 being the worst imaginable pain possible. The epidural steroid injection group is compared to the gabapentin group.
Time Frame: 3 months from the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Gabapentin Group: This group received gabapentin and a placebo intramuscular injection.
- Epidural Steroid: This group received an epidural steroid injection and placebo gabapentin.
Arm/Group | Gabapentin Group | Epidural Steroid
Number analyzed (Participants) | 72 | 73
units on a scale | 3.7 (2.8) | 3.4 (2.7)

3. Primary Outcome: Worst Leg Pain at 1 Month Measured Using the Numeric Pain Scale
Description: as for outcome 1
Time Frame: 1 month from the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 73 | 72
units on a scale | 4.9 (3.1) | 5.8 (3.0)

4. Primary Outcome: Worst Leg Pain at 3 Months Measured Using the Numeric Pain Scale
Description: This outcome measure compares the worst leg pain at baseline to the worst leg pain at 3 months after the start of treatment. This is measured using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0-10. 0 being no pain at all and 10 being the worst imaginable pain possible. The epidural steroid injection group is compared to the gabapentin group.
Time Frame: 3 months from the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 73 | 72
units on a scale | 5.2 (3.4) | 5.5 (3.4)

5. Secondary Outcome: Average Back Pain at 1 Month Measured Using the Numeric Pain Scale
Description: This outcome measure compares the average back pain at baseline to the average back pain 1 month after the start of treatment. This is measured using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0-10. 0 being no pain at all and 10 being the worst imaginable pain possible. The epidural steroid injection group is compared to the gabapentin group.
Time Frame: 1 month fromt he start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 73 | 72
units on a scale | 3.5 (2.6) | 3.6 (2.6)

6. Secondary Outcome: Average Back Pain at 3 Months Measured Using the Numeric Pain Scale
Description: This outcome measure compares the average back pain at baseline to the average back pain at 3 months after the start of treatment. This is measured using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0-10. 0 being no pain at all and 10 being the worst imaginable pain possible. The epidural steroid injection group is compared to the gabapentin group.
Time Frame: 3 months from the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 73 | 72
units on a scale | 3.9 (2.7) | 3.7 (2.5)

7. Secondary Outcome: Outcomes Related to Disability Measured at 1 Month Using the Oswestry Disability Index
Description: Functional capacity measured using Oswestry disability index. The range of possible scores for Oswestry Disability Index are 0-100. 0 is equated with no disability and 100 is the maximum disability possible.
Time Frame: 1 month after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 73 | 72
units on a scale | 32.6 (18.3) | 29.6 (16.0)

8. Secondary Outcome: Outcomes Related to Disability Measured at 3 Month Using the Oswestry Disability Index
Description: as for outcome 7
Time Frame: 3 months after the start of treatment
Measure: Mean (Standard Deviation); unit: participants
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 73 | 72
participants | 33.6 (19.4) | 29.6 (16.3)

9. Secondary Outcome: Global Perceived Effect of Treatment at 3 Months After the Start of Treatment
Description: The participant is asked "Are you satisfied with the treatment you have received so far? Participants could respond yes or no. This is measured 3 months after the start of treatment.
Time Frame: 3 months after the start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 73 | 72
Participants
  Yes | 27 | 21
  No | 46 | 51

10. Secondary Outcome: Global Perceived Effect of Treatment at 1 Month After the Start of Treatment
Description: The participant is asked "Are you satisfied with the treatment you have received so far? Participants could respond yes or no. This is measured 1 month after the start of treatment.
Time Frame: 1 month after the start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 73 | 72
Participants
  Yes | 48 | 33
  No | 25 | 39

11. Secondary Outcome: Worst Back Pain at 1 Month Measured Using the Numeric Pain Scale
Description: This outcome measure compares the worst back pain at baseline to the worst back pain at 1 months after the start of treatment. This is measured using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0-10. 0 being no pain at all and 10 being the worst imaginable pain possible. The epidural steroid injection group is compared to the gabapentin group.
Time Frame: 1 month from the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 73 | 72
units on a scale | 5.1 (2.9) | 5.4 (3.2)

12. Secondary Outcome: Worst Back Pain at 3 Months Measured Using the Numeric Pain Scale
Description: This outcome measure compares the worst back pain at baseline to the worst back pain at 3 months after the start of treatment. This is measured using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0-10. 0 being no pain at all and 10 being the worst imaginable pain possible. The epidural steroid injection group is compared to the gabapentin group.
Time Frame: 3 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 73 | 72
units on a scale | 5.6 (3.2) | 5.6 (3.1)

13. Secondary Outcome: Proceeded to Surgery Within Year of Enrollment
Description: This is a measure of participants that proceeded to surgery within a year of enrollment
Time Frame: Measured within the year of enrollment in the study
Population: Data for this outcome measure was collected one year following the last follow-up. Data was not available for one participant in the epidural steroid injection arm and for three in the gabapentin arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Steroid Injection | Gabapentin
Number analyzed (Participants) | 72 | 69
Participants | 9 | 10

ADVERSE EVENTS:
Arm/Group | Epidural Steroids | Gabapentin
Serious Adverse Events (participants affected / at risk) | 15/73 | 19/72
Other Adverse Events (participants affected / at risk) | 24/73 | 26/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural Steroids (N=73) | Gabapentin (N=72)
Excessive pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) — Excessive pain after epidural steroid injection or intramuscular injection
Fever or infection (Infections and infestations) | 2 (2) | 0 (0) — Those who experienced fever or infection after epidural steroid injection or intramuscular placebo injection.
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Fall after procedure
Vasovagal (Cardiac disorders) | 0 (0) | 2 (2)
Coginitve (Nervous system disorders) | 5 (5) | 7 (7) — Decrease cognition
Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Swelling (Immune system disorders) | 0 (0) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1) | 2 (2)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural Steroids (N=73) | Gabapentin (N=72)
Gastrointestinal Upset (Gastrointestinal disorders) | 13 (13) | 8 (8)
Weight Gain (Metabolism and nutrition disorders) | 4 (4) | 7 (7)
Sedation Fatigue (Nervous system disorders) | 7 (7) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes